CLINICAL TRIAL: NCT01881217
Title: An Open-label, Phase I, Dose-escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous BAY 1179470 in Subjects With Advanced, Refractory Solid Tumors.
Brief Title: First-in-man Dose Escalation Study of BAY1179470 in Patients With Advanced, Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16182
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Neoplasms
Keywords: Phase I; Dose escalation; Advanced, refractory solid tumors; FGFR2
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BAY1179470 (Dose escalation) (Experimental): BAY1179470 will be administered as a 1-hour intravenous infusion every 21 days.
  Interventions: Drug: BAY1179470
- BAY1179470 (additional) (Experimental): Additional cohort: BAY1179470 will be administered as a 1-hour intravenous infusion every 21 days.
  Interventions: Drug: BAY1179470
- BAY1179470 (expansion) (Experimental): Expansion cohort: BAY1179470 will be administered as a 1-hour intravenous infusion every 21 days.
  Interventions: Drug: BAY1179470

INTERVENTIONS:
Drug: BAY1179470 — BAY1179470 will be administered as a 1-hour intravenous infusion.

SUMMARY:
An open-label, non-randomized, Phase I dose-escalation study designed to assess the safety, tolerability, pharmacokinetics(PK) /pharmacodynamics( PD) and tumor response profile of BAY1179470 in subjects with advanced, refractory solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced, histologically or cytologically confirmed solid tumors refractory to any standard therapy or have no standard therapy available or subjects actively refuse any treatment which would be regarded standard
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1 and a life expectancy of at least 3 months
* Adequate bone marrow, liver, and renal function.

For subjects in the additional cohort:

* Subjects with advanced, histologically or cytologically confirmed gastric cancer.
* At least moderate FGFR2 expression in the tumor tissue from archival samples is confirmed

Exclusion Criteria:

* History of severe allergic reactions to monoclonal antibody therapy
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 90 mmHg, despite optimal medical management
* Any condition that is unstable or could jeopardize the safety of the subject and his / her compliance in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-06-28 (Actual); Primary Completion 2016-03-18 (Actual); Study Completion 2016-08-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a Measure of Safety and Tolerability | Up to 2 years
Maximum drug concentration versus time curve (AUC) from zero to infinity after single (first) and multiple doses of BAY1179470 | Cycle 1 and 2: pre-dose, 0.5, 1 , 2, 3, 5, 8, 24, 48, 72, 168 and 336 hours after start of the infusion, Cycle 3 and 4: pre-dose and 1 hour after start of the infusion; each cycle is 21 days
Maximum drug concentration (Cmax) and minimal drug concentration (Cmin) of BAY1179470 in plasma after single and multiple dose administration | Cycle 1 and 2: pre-dose, 0.5, 1 , 2, 3, 5, 8, 24, 48, 72, 168 and 336 hours after start of the infusion, Cycle 3 and 4: pre-dose and 1 hour after start of the infusion; each cycle is 21 days

SECONDARY OUTCOMES:
Tumor response | Every 42 days
  Tumor response will be evaluated based on the RECIST (Response Evaluation Criteria in Solid Tumors) 1.1 criteria.
Biomarker (plasma) | Cycle 1: pre-dose, 24 hours after start of the infusion and Day 15, Cycle 2, 3 and 4: pre-dose; each cycle is 21 days
Biomarker (biopsy) | Cycle 1: pre-dose and Day 8; cycle 1 is 21 days
  Additional cohort only
Immunogenicity | Cycle 1 and Cycle 2 pre-dose and every second cycle thereafter pre-dose. End of treatment visit and follow-up visit up to 2 years; each cycle is 21 days
  Analyzed for anti-BAY 1179470 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- Japan (5):
  - Kashiwa, Chiba
  - Kita-Adachigun, Saitama
  - Chuo-ku, Tokyo
  - Koto-ku, Tokyo
  - Fukuoka
- Singapore, Singapore
- Seoul, South Korea